CLINICAL TRIAL: NCT00235924
Title: Study Assessing the Effects on Endometrium and Breast of a Standardized Isoflavone Extract(Phytosoya) in Post Menopausal Women.
Brief Title: Study Assessing the Effects on Endometrium and Breast of Isoflavone in Post Menopausal Women
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laboratoires Arkopharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHY04GE01
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2005-12-08 (Estimated); Status verified 2005-10

CONDITIONS: Postmenopause
Keywords: menopause; isoflavone; endometrial safety; breast innocuity assessment; hot flushes
MeSH Terms: conditions — Hot Flashes | interventions — Soybean Proteins

INTERVENTIONS:
Drug: soy isoflavone

SUMMARY:
The main objective of this study is to determine the effects on the endometrium and breast of 70 mg daily dose of isoflavones.

DETAILED DESCRIPTION:
This is an international multicentre open study, assessing the innocuity on breast and endometrium of a 70 mg daily dose of isoflavones standardized extract (Phytosoya).

This study follows the European guidelines :one-year treatment duration, biopsy and mammography performed at the beginning and at the end of the trial, recruitment of enough subjects in order to have 300 patients with an evaluable biopsy after one year of treatment.

After 3 weeks of screening phase, the patients will be taken Phytosoya during 52 weeks. At the end of the first year of treatment, an endometrial biopsy, an endovaginal ultrasonography, a mammography, breast ultrasounds, a clinical examination and a biological assessment will be performed.

In addition, it will be proposed to patients to continue treatment during 2 additional years. At the end of the third year,the same examinations will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Not hysterectomised women
* Post menopausal (at least 2 years)
* FSH superior to 30 UI/l and oestradiol inferior to 35 ng/ml
* Presenting with hot flushes (but not incapacitating) or climacteric symptoms

Exclusion Criteria:

* History of endometrial hyperplasia
* Known hormono-dependent malignant tumours
* BMI superior to 30 Kg/m2
* Uncontrolled arterial hypertension
* Known renal or liver insufficiency
* Recent or evolutive thromboembolic disease
* Unexplained bleeding, endometrial polyps, submucous myomas, active endometriosis, ovarian cyst superior to 30 mm
* Local hormonal treatment, raloxifene,tibolone within the 3 months before V1 and during the study
* HRT and DHEA within the 3 months before V2 and during the study
* isoflavones within the 2 months before V2 and during the study
* clonidine, beta-alanine, veralipride within 1 month before V1 and during the study.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-06

PRIMARY OUTCOMES:
- Endometrial innocuity (endometrial biopsy result)

SECONDARY OUTCOMES:
- Mammary innocuity (mammography results)
- climacteric symptoms
-Lipid profile
-gynaecological and general safety

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MARES, Professor, Study Chair — Hospital of Caremeau, Nîmes, FRANCE; Santiago PALACIOS, Professor, Principal Investigator — Instituto Palacios, Madrid, SPAIN; Bruno PORNEL, Doctor, Principal Investigator — Brussels Menopause Center, Bruxelles, BELGIUM; John EDEN, Professor, Principal Investigator — Sydney Menopause Center, Sydney, AUSTRALIA